CLINICAL TRIAL: NCT01510587
Title: Family Influences to Prevent Childhood Obesity: An Integrated Research and Outreach Program for Parents of Montana 4-H Youth
Brief Title: Family Influences to Prevent Childhood Obesity
Acronym: 4-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wesley Lynch, Professor of Psychology, Montana State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4W3685; 2009-55215-05334 (Other Grant/Funding Number: USDA-NIFA-AFRI)
Record Dates: First submitted 2012-01-07; First posted 2012-01-16 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Childhood Obesity
Keywords: obesity; prevention; preteen; nutrition; physical activity; body image; family dynamics
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4-Health Educational curriculum (Experimental): Parents participate in 10 face-to-face educational sessions delivered by Extension Agents at individual county locations over a 8-month period (fall to spring).
  Interventions: Behavioral: 4-Health Educational curriculum
- Healthy Living Information (Active Comparator): Participants receive 10 mailed packets of written information derived from USDA's MyPlate website on approximately the same schedule as meetings of the experimental group.
  Interventions: Behavioral: Healthy Living Information

INTERVENTIONS:
Behavioral: 4-Health Educational curriculum — During the intervention, parents meet about every 3 weeks (90 min/session) in small groups with facilitators. During meetings classroom activities aim to integrate 3 areas: 1) parents' knowledge about healthy diets, physical activity and improved body image; 2) parents' understanding, skills and potential roles as positive change-agents (i.e., parenting and behavior management); and 3) parents' learning and practicing cognitive-behavioral exercises that encourage specific skills within the family/home setting. Between monthly meetings, participants explore a suggested online websites or facilitator-assigned questions and provide feedback. The majority of outside time/assignments for parents is spent doing take-home activities with their preteen child and family.
  Other Names: 4-Health Educational Program
  Arms: 4-Health Educational curriculum
Behavioral: Healthy Living Information — During the Healthy Living Information intervention, participants receive packets delivered to their homes by mail at intervals similar to the meeting intervals for the educational curriculum intervention. (10 total packets.) Approximately every three weeks between late September 2011 and April 2012, corresponding approximately to the meeting times for the 4-Health Educational Program, participants in the Healthy Living Information control group receive mailed packets of information.
  Arms: Healthy Living Information

SUMMARY:
The main goal of this project is to develop, deliver, and assess the efficacy of a parent-centered educational program (4-Health) designed to prevent preteen children from becoming overweight.

DETAILED DESCRIPTION:
Previous studies suggest that parents can play a key role in preventing childhood obesity. Program objectives are to increase parents' knowledge and skills related to nutrition, physical activity, and best parenting practices. Developed from a successful existing program, the proposed program will include a novel classroom curriculum coupled with outside exercises, online resources, and a strong social support network. The curriculum will be developed with input from stakeholders during year 1 and implemented during years 2 and 3. The target groups are children and parents participating in 4-H Youth Development Programs in Montana. Intervention effectiveness will be assessed by comparing objective and self-report data between-groups (intervention vs. control) and within-groups (pre- to post-intervention and at 6 month follow-up). Physiological measures, including resting heart rate, blood pressure, body weight and age- and gender-specific BMI z-scores of children, are expected to show significant improvement among children of parents receiving the intervention compared to a mailed written materials control group. In addition, positive changes are anticipated in outcome measures provided by parents and children, including levels of daily physical activity and specific food and nutrition behaviors. Positive changes in parents' attitudes about diet, body image, and their perceived feeding practices before versus after intervention and at 6 month follow-up are also expected. This project will lead to improved understanding of how parents influence child obesity and improved interventions to prevent obesity.

ELIGIBILITY:
Inclusion Criteria:

* Parent of 8-12 year old child in 4-H Youth Development Programs in Montana
* Child of parent enrolled in study

Exclusion Criteria:

* Parent of child age outside the 8-12 year old range at start of trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change child body mass index z-score. | Baseline, end of program, 6 month follow up

SECONDARY OUTCOMES:
Change in youth and parent self-reported physical activity. | Baseline, end of program, 6 month follow up
Change in child and parent physical activity self-efficacy. | Baseline, end of program, 6 month follow up
Change in child and parent dietary self-efficacy. | Baseline, end of program, 6 month follow up
Change in child and parent body image. | Baseline, end of program, 6 month follow up
Change in child quality of life via self-report and parent report. | Baseline, end of program, 6 month follow up
Change in parent body mass index. | Baseline, end of program, 6 month follow up
Change in child and parent diastolic and systolic blood pressure. | Baseline, end of program, 6 month follow up
Change in child and parent heart rate. | Baseline, end of program, 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Lynch, PhD, Principal Investigator — Montana State University; Lynn Paul, PhD, RD, Principal Investigator — Montana State University; Jill Martz, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

REFERENCES:
- [Derived] Lynch WC, Martz J, Eldridge G, Bailey SJ, Benke C, Paul L. Childhood obesity prevention in rural settings: background, rationale, and study design of '4-Health,' a parent-only intervention. BMC Public Health. 2012 Apr 2;12:255. doi: 10.1186/1471-2458-12-255. PMID 22471650